CLINICAL TRIAL: NCT04416945
Title: Targeting High-risk Populations With Enhanced Reactive Case Detection: a Study to Assess the Effectiveness and Feasibility for Reducing Plasmodium Falciparum and P. Vivax Malaria in Southern Lao Peoples Democratic Republic
Brief Title: Targeting High Risk Populations With Enhanced Reactive Case Detection in Southern Lao Peoples Democratic Republic
Acronym: COMBAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, San Francisco (Other)
Collaborators: Center for Malariology, Parasitology, and Entomology (Unknown); Tulane University School of Public Health and Tropical Medicine (Other); University of Massachusetts, Amherst (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: 19-27966
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Plasmodium Falciparum Malaria; Plasmodium Vivax Malaria
MeSH Terms: conditions — Malaria, Falciparum; Malaria, Vivax | interventions — Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RACD (Experimental): Reactive case detection led by VMWs in response to cases in study area HCCA, with follow up testing with HS-RDTs/RDTs in both villages and forest workers; referrals for qualitative G6PD testing for P. vivax cases and 14-day PQ for G6PD non-deficient
  Interventions: Other: Household Reactive Case Detection; Other: RACD of cases' co-workers/co-travelers; Other: Case Management and Follow-up
- Control (Active Comparator): Standard of care including case management through health facilities and malaria posts/VMWs; village-based RACD conducted by district staff in some areas
  Interventions: Other: Case Management and Follow-up

INTERVENTIONS:
Other: Household Reactive Case Detection — Within 7 days of the index case notification, all members of the index case's household and everyone in the neighboring five households will then be invited to participate in the study. After consenting, a finger stick blood sample will be collected for each consenting individual for testing with the HS-RDT for P. falciparum, a standard combination RDT, and four blood spots on filter paper.
  Arms: RACD
Other: RACD of cases' co-workers/co-travelers — Index cases will be screened by the VMW at their households at the time of case investigation to determine if they have traveled or worked in a forest or forest-fringe area within the past 30 days. If eligible, the case will trigger two reactive recruitment strategies to screen and treat others who recently traveled or worked with the case in a forest or forest-fringe location:
  1. Peer-referral RACD (PR-RACD): In this strategy, the case will identify specific co-travelers or co-workers resident in their village who had spent the night with the case at a forest or forest-fringe area and spent the night there in the past 30 days.
  2. Venue-based RACD (VB-RACD): In this strategy, co-workers will be recruited directly from (accessible) forest or forest-fringe work sites where the index case worked and spent at least one night in the past 30 days.
  Arms: RACD
Other: Case Management and Follow-up — All individuals who test positive by either HS-RDT or Standard RDT will be told of their results and treated on site per national guidelines:
  * Individuals with P. falciparum infection will be treated with an age-appropriate course of artemether-lumefantrine (AL) and a single low dose of primaquine (SLD-PQ). Weight-based dosing is described in Tables 2 and 3 below.
  * At all study sites in Lao Peoples Democratic Republic, patients with a P. vivax infection identified by RDT (both febrile and asymptomatic) will be given a unique coded and signed informational letter directing them to the nearest district hospital (or other testing facility) for G6PD deficiency testing and possible radical cure administration depending on results. At the health facility, G6PD normal individuals will be treated with AL and a 14-day course of PQ, whereas G6PD deficient individuals will receive AL alone as per the national guidelines and referred to a hospital for further primaquine management decisions.

SUMMARY:
This study assesses the effectiveness and feasibility of enhanced reactive case detection (RACD) targeting high-risk villages and forest workers for reducing Plasmodium falciparum and Plasmodium vivax transmission in southern Lao Peoples Democratic Republic. The authors hypothesize that enhanced community-based RACD will be more effective than standard of care case management and RACD at reducing P. falciparum and P. vivax confirmed case incidence and parasite prevalence over an 18-month period in Lao Peoples Democratic Republic.

DETAILED DESCRIPTION:
In the Greater Mekong Subregion (GMS), the risk of malaria infection is often due not to village-based transmission but rather to occupational and behavioral risk factors leading to exposure in forest settings. Additionally, a substantial portion of infections are asymptomatic and/or submicroscopic, limiting the scope of current diagnostics and surveillance approaches. The proposed research will evaluate the effectiveness of reactive case detection (RACD) using highly-sensitive rapid diagnostic tests (HS-RDTs), targeting both village and forest working populations, compared to control for reducing the health center catchment-level incidence and prevalence of P. falciparum and P. vivax within two provinces in Lao People's Democratic Republic.

To test this hypothesis, this study will employ a cluster randomized controlled trial design with two comparison arms: (1) Control: standard of care - passive case management provided through community-based Village Malaria Workers (VMWs) and existing health facilities; includes village-based RACD with conventional rapid diagnostic tests (RDTs) conducted by district surveillance teams and (2) enhanced community-based RACD: RACD conducted by community-based VMWs using both HS-RDTs and conventional RDTs within villages and among forest workers.

The primary outcome measures to assess effectiveness include P. falciparum and P. vivax confirmed case incidence over the study period; PCR-based P. falciparum and P. vivax prevalence at end line; and HS-RDT test positivity rate in village and forest worker RACD. Secondary outcomes measures will examine the operational feasibility, safety, and acceptability of VMW-led reactive approaches and glucose-6-phosphate dehydrogenase (G6PD) testing, referral to district or provincial-level facilities, safety and treatment adherence for P. vivax cases.

ELIGIBILITY:
RACD:

- Inclusion Criteria

* Inclusion Criteria for index cases: Presented as a confirmed malaria case to an intervention health facility or village malaria worker, and lives in a village within a selected intervention health facility catchment area, or worked or spent at least one night at a forest or forest-fringe site in the past 30 days located within an intervention health facility catchment area
* Inclusion criteria for village residents: Lives in a village within a selected intervention health facility catchment area and in one of the five households closest to the residence of an index case of malaria
* Inclusion criteria for co-worker/traveler referral: Worked or traveled and spent at least one night in forest in past 30 days in same location within an intervention health facility catchment area as an index case of malaria
* Inclusion criteria for all participants: Willing and available to participate in the study

Informed consent for participant under the age of 18 will be provided by the parent or guardian.

- Exclusion Criteria:

* Previous participation in the study as a result of any RACD event in the past 30 days.
* Individuals with suspected severe malaria or other severe illness (including those with symptoms of severe anemia, prostration, impaired consciousness, respiratory distress, convulsions, circulatory collapse, abnormal bleeding, jaundice or passing dark urine) will be excluded from the treatment component and referred to the nearest health facility for clinical assessment and treatment

Min Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 31443 (Estimated)
Dates: Start 2020-09-20 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Confirmed P. falciparum and P. vivax malaria parasite incidence | 4 months
  This is defined as the number of outpatient (OPD) malaria confirmed and suspected cases per person per year for each Health Center Catchment Area (HCCA), as ascertained from the health facility registers, utilizing administrative catchment population size estimates for the exposure denominator.
PCR-based P. falciparum and P. vivax parasite prevalence in sampled HCCAs | 4 months
  This is defined as the proportion of individuals ≥18 months old with P. falciparum or P. vivax infection (detected by PCR) out of all individuals ≥18 months tested within the end line survey (2020).
HS-RDT/RDT-based test positivity rate in village and forest-based reactive case detection | 4 months
  This is defined as the proportion of all individuals tested by HS-RDT/RDT in response to an index cases, with a positive HS-RDT/RDT, among the population older than 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Bennett, MA, PhD, Principal Investigator — University of California, San Francisco; Viengxay Vanisaveth, MD, Principal Investigator — Center of Malariology, Parasitology, Entomology in Laos
Locations (1):
- Center for Malariology, Parasitology, Entomology, Laos Ministry of Health, Vientiane, Laos

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with any parties outside of the study team.

REFERENCES:
- [Background] Bousema T, Griffin JT, Sauerwein RW, Smith DL, Churcher TS, Takken W, Ghani A, Drakeley C, Gosling R. Hitting hotspots: spatial targeting of malaria for control and elimination. PLoS Med. 2012 Jan;9(1):e1001165. doi: 10.1371/journal.pmed.1001165. Epub 2012 Jan 31. PMID 22303287
- [Background] Cotter C, Sturrock HJ, Hsiang MS, Liu J, Phillips AA, Hwang J, Gueye CS, Fullman N, Gosling RD, Feachem RG. The changing epidemiology of malaria elimination: new strategies for new challenges. Lancet. 2013 Sep 7;382(9895):900-11. doi: 10.1016/S0140-6736(13)60310-4. Epub 2013 Apr 15. PMID 23594387
- [Background] Moonen B, Cohen JM, Snow RW, Slutsker L, Drakeley C, Smith DL, Abeyasinghe RR, Rodriguez MH, Maharaj R, Tanner M, Targett G. Operational strategies to achieve and maintain malaria elimination. Lancet. 2010 Nov 6;376(9752):1592-603. doi: 10.1016/S0140-6736(10)61269-X. Epub 2010 Oct 28. PMID 21035841
- [Background] Hustedt J, Canavati SE, Rang C, Ashton RA, Khim N, Berne L, Kim S, Sovannaroth S, Ly P, Menard D, Cox J, Meek S, Roca-Feltrer A. Reactive case-detection of malaria in Pailin Province, Western Cambodia: lessons from a year-long evaluation in a pre-elimination setting. Malar J. 2016 Mar 1;15:132. doi: 10.1186/s12936-016-1191-z. PMID 26931488
- [Background] Rossi G, Van den Bergh R, Nguon C, Debackere M, Vernaeve L, Khim N, Kim S, Menard D, De Smet M, Kindermans JM. Adapting Reactive Case Detection Strategies for falciparum Malaria in a Low-Transmission Area in Cambodia. Clin Infect Dis. 2018 Jan 6;66(2):296-298. doi: 10.1093/cid/cix781. PMID 29020325
- [Background] Das S, Peck RB, Barney R, Jang IK, Kahn M, Zhu M, Domingo GJ. Correction to: Performance of an ultra-sensitive Plasmodium falciparum HRP2-based rapid diagnostic test with recombinant HRP2, culture parasites, and archived whole blood samples. Malar J. 2019 Feb 4;18(1):33. doi: 10.1186/s12936-019-2669-2. PMID 30717748
- [Background] Landier J, Parker DM, Thu AM, Lwin KM, Delmas G, Nosten FH; Malaria Elimination Task Force Group. Effect of generalised access to early diagnosis and treatment and targeted mass drug administration on Plasmodium falciparum malaria in Eastern Myanmar: an observational study of a regional elimination programme. Lancet. 2018 May 12;391(10133):1916-1926. doi: 10.1016/S0140-6736(18)30792-X. Epub 2018 Apr 24. PMID 29703425
- [Background] Howes RE, Dewi M, Piel FB, Monteiro WM, Battle KE, Messina JP, Sakuntabhai A, Satyagraha AW, Williams TN, Baird JK, Hay SI. Spatial distribution of G6PD deficiency variants across malaria-endemic regions. Malar J. 2013 Nov 15;12:418. doi: 10.1186/1475-2875-12-418. PMID 24228846
- [Background] White MT, Karl S, Battle KE, Hay SI, Mueller I, Ghani AC. Modelling the contribution of the hypnozoite reservoir to Plasmodium vivax transmission. Elife. 2014 Nov 18;3:e04692. doi: 10.7554/eLife.04692. PMID 25406065
- [Background] Douglas NM, Poespoprodjo JR, Patriani D, Malloy MJ, Kenangalem E, Sugiarto P, Simpson JA, Soenarto Y, Anstey NM, Price RN. Unsupervised primaquine for the treatment of Plasmodium vivax malaria relapses in southern Papua: A hospital-based cohort study. PLoS Med. 2017 Aug 29;14(8):e1002379. doi: 10.1371/journal.pmed.1002379. eCollection 2017 Aug. PMID 28850568
- [Background] Ministry of Health Lao PDR. The Evaluation of G6PD Rapid Tests and the Use of Primaquine for the Treatment of Plasmodium Vivax Infections in Luangprabang, Savannakhet and Champasak Provinces (Apr-Nov 2015). (2015).
- [Background] Center for Malariology Parasitology and Entomology Lao PDR. Lao PDR Malaria National Strategic Plan 2016-2020. (2015).
- [Background] WHO. Updated WHO policy recommendation: Single dose primaquine as a gametocytocide in Plasmodium falciparum malaria. World Health Organisation (2012).
- [Background] Baum E, Sattabongkot J, Sirichaisinthop J, Kiattibutr K, Davies DH, Jain A, Lo E, Lee MC, Randall AZ, Molina DM, Liang X, Cui L, Felgner PL, Yan G. Submicroscopic and asymptomatic Plasmodium falciparum and Plasmodium vivax infections are common in western Thailand - molecular and serological evidence. Malar J. 2015 Feb 25;14:95. doi: 10.1186/s12936-015-0611-9. PMID 25849211
- [Background] Corran P, Coleman P, Riley E, Drakeley C. Serology: a robust indicator of malaria transmission intensity? Trends Parasitol. 2007 Dec;23(12):575-82. doi: 10.1016/j.pt.2007.08.023. Epub 2007 Nov 7. PMID 17988945
- [Background] Chan CW, Sakihama N, Tachibana S, Idris ZM, Lum JK, Tanabe K, Kaneko A. Plasmodium vivax and Plasmodium falciparum at the crossroads of exchange among islands in Vanuatu: implications for malaria elimination strategies. PLoS One. 2015 Mar 20;10(3):e0119475. doi: 10.1371/journal.pone.0119475. eCollection 2015. PMID 25793260
- [Background] Beutler E, Duparc S; G6PD Deficiency Working Group. Glucose-6-phosphate dehydrogenase deficiency and antimalarial drug development. Am J Trop Med Hyg. 2007 Oct;77(4):779-89. PMID 17978087
- [Background] Campbell MK, Piaggio G, Elbourne DR, Altman DG; CONSORT Group. Consort 2010 statement: extension to cluster randomised trials. BMJ. 2012 Sep 4;345:e5661. doi: 10.1136/bmj.e5661. No abstract available. PMID 22951546

DOCUMENTS (1):
  • Study Protocol (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/45/NCT04416945/Prot_000.pdf